CLINICAL TRIAL: NCT02984605
Title: Effects of Nutrition Meal Replacement and Individualized Exercise Prescription on Metabolism in Overweight and Obese Type 2 Diabetes
Brief Title: Effects of Nutrition Meal Replacement and Individualized Exercise Prescription on Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai University of Sports National Science Park (Unknown); Yinhang Community Health Service Center of Yangpu District (Unknown); Dinghai Community Health Service Center of Yangpu District (Unknown); Kongjiang Community Health Service Center of Yangpu District (Unknown); Daqiao Community Health Service Center of Yangpu District (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-046
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Overweight; Obesity; Type2 Diabetes
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional group (Experimental): Arm：Hypoglycemic agents + Nutrition meal replacement & exercise prescription
  Hypoglycemic agents in combined with 1 times a day with bags of nutritional meal replacement and exercise
  Interventions: Dietary Supplement: nutritional meal replacement
- Control group (No Intervention): Arm：Hypoglycemic agents
  without take nutrition meal replacement & exercise prescription

INTERVENTIONS:
Dietary Supplement: nutritional meal replacement — 1 times a day with bags of nutritional meal replacement + individualized exercise prescription
  Arms: Interventional group

SUMMARY:
This study evaluates the nutritional meal replacement and individualized exercise prescription intervention on overweight and obese type 2 diabetes mellitus. Half of participants will receive nutritional meal replacement and individualized exercise prescription on the basis of conventional glucose-lowering treatment, while the other half will only receive conventional glucose-lowering treatment.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic metabolic disease which seriously threatens people's health at present. Although new drugs for the treatment of diabetes continue to emerge, but the effect of diabetes treatment is still not satisfactory. Medical nutrition therapy (nutrition therapy medical, MNT) and exercise therapy are essential measures for prevention and control of diabetes at any stage of the natural course of the disease, especially for the overweight and obese patients with type 2 diabetes. However, at present, the majority of patients could not get the guide from nutrition specialist and sports specialist. In addition, the existing diet programs are often more complex, difficult to implement and adhere to in daily life, and exercise programs are often lack of targeted. In view of this, the Shanghai peak Sports Management Co., Ltd. developed a kind of nutritional meal replacement for weight loss. The nutritional powder has the characteristics of high nutrition, low calorie, low glycemic and strong satiety, and the heat is only 126kcal, and have a good sense of satiety. Studies have shown that 1 times a day with bags of nutritional meal replacement instead of 1 meals for obese people have a role in weight loss. In theory, the meal is also suitable for diabetes patients, especially overweight and obese type 2 diabetes, such as the combination of individual exercise prescription may be better, but there is still a lack of relevant research. In view of this, we proposed a joint sports workers, explore nutritional and individualized exercise prescription intervention on overweight and obese type 2 diabetes mellitus, to explore suitable for China's diabetes lifestyle intervention measures, improve the level of prevention and treatment of diabetes in China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of overweight and obesity type 2 diabetes
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, MD, Principal Investigator — YinXing Community Health Service Center of Yangpu District; Wenbin Liu, MD, Principal Investigator — Dinghai Community Health Service Center of Yangpu District; Xiaoyi Che, MD, Principal Investigator — Kongjiang Community Health Service Center of Yangpu District; Hui Liu, MD, Principal Investigator — Daqiao Community Health Service Center of Yangpu District

IPD SHARING:
Plan to Share IPD: No